CLINICAL TRIAL: NCT05165823
Title: The Significance of Sodium Balance for Blood Pressure in Patients With Essential Hypertension and the Value of Salt-blood Test in Identifying Salt Sensitive Patients With Hypertension
Brief Title: The Significance of Sodium Balance and the Value of Salt-blood Test in Identifying Salt Sensitive Patients
Acronym: VASA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Camilla Lundgreen Duus, Doctor, Ph.D.-student, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLD-2-2021
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Hypertension,Essential
Keywords: Salt sensitivity; Sodium sensitivity; Salt restriction; Salt-blood test; Dietary intervention; Hypertension
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium restriction (Experimental)
  Interventions: Behavioral: Sodium restriction
- Usual diet (No Intervention)

INTERVENTIONS:
Behavioral: Sodium restriction — Participants will be guided in minimizing sodium intake. Guidance will be both oral and written. Bread with low sodium content will be offered to the participants.
  Arms: Sodium restriction

SUMMARY:
This is a randomized controlled trial with 72 patients with hypertension examining the effects on blood pressure of sodium restriction and whether the blood analysis Salt-blood test is associated to a decrease in blood pressure. Patients will be randomized 2:1 to either sodium restriction or usual diet for 4 weeks. Baseline measures will be done before intervention and outcome measures after the 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≤ 35 kg/m2
* Essential hypertension
* eGFR > 15 ml/min/1,73m2
* Albumine-to-creatinine-ratio < 500 mg/g
* Safe anticonception if women in childbearing age.
* Able to adhere to dietary regimen

Exclusion Criteria:

* Secondary hypertension
* Clinically significant heart failure (NYHA 3-4)
* Clinically significant liver disease
* Diabetes mellitus (type 1 and 2)
* Active cancer (except skin cancer)
* Renal transplant
* Recent stroke, transcient ischemic attack or myocardial infarction (within 6 months)
* Proliferative glomerulonephritis or ANCA-related disease
* Continuous immunosuppressant treatment
* Pregnancy or lactation
* Alcohol abuse
* If the investigator finds the participant unfit to complete the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Change in systolic 24-hour blood pressure | Measured before and after 4 weeks' intervention
  Difference in systolic blood pressure measured before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Lundgreen Duus, Principal Investigator — University Clinic in Nephrology and Hypertension
Locations (1):
- University Clinic in Nephrology and Hypertension, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duus CL, Nielsen SF, Hornstrup BG, Mose FH, Bech JN. Self-Performed Dietary Sodium Reduction and Blood Pressure in Patients With Essential Hypertension: A Randomized Clinical Trial. J Am Heart Assoc. 2024 Jun 18;13(12):e034632. doi: 10.1161/JAHA.124.034632. Epub 2024 Jun 6. PMID 38842286